CLINICAL TRIAL: NCT05740813
Title: HEALEY ALS Platform Trial - Regimen F ABBV-CLS-7262
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Merit E. Cudkowicz, MD (Other)
Collaborators: Calico Life Sciences LLC (Industry)
Responsible Party: Sponsor-Investigator, Merit E. Cudkowicz, MD, Chief, Neurology Department, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019P003518F
Record Dates: First submitted 2023-02-12; First posted 2023-02-23 (Actual); Results first posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; Placebo-Controlled; Double-Blind; Regimen Specific Appendix; Lou Gehrig's Disease; ABBV-CLS-7262; Calico Life Sciences
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ABBV-CLS-7262 Dose 1 (Experimental)
  Interventions: Drug: ABBV-CLS-7262 Dose 1
- ABBV-CLS-7262 Dose 2 (Experimental)
  Interventions: Drug: ABBV-CLS-7262 Dose 2
- Matching Placebo (Placebo Comparator)
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: ABBV-CLS-7262 Dose 1 — ABBV-CLS-7262 is administered orally once per day for 24 weeks.
  Arms: ABBV-CLS-7262 Dose 1
Drug: ABBV-CLS-7262 Dose 2 — ABBV-CLS-7262 is administered orally once per day for 24 weeks.
  Arms: ABBV-CLS-7262 Dose 2
Drug: Matching Placebo — Matching placebo is administered orally once per day for 24 weeks.
  Arms: Matching Placebo

SUMMARY:
The HEALEY ALS Platform Trial is a perpetual multi-center, multi-regimen clinical trial evaluating the safety and efficacy of investigational products for the treatment of ALS.

Regimen F will evaluate the safety and efficacy of a single study drug, ABBV-CLS-7262, in participants with ALS.

DETAILED DESCRIPTION:
The HEALEY ALS Platform Trial is a perpetual multi-center, multi-regimen clinical trial evaluating the safety and efficacy of investigational products for the treatment of ALS. This trial is designed as a perpetual platform trial. This means that there is a single Master Protocol dictating the conduct of the trial. The HEALEY ALS Platform Trial Master Protocol is registered as NCT04297683. Once a participant enrolls into the Master Protocol and meets all eligibility criteria, the participant will be eligible to be randomized into any currently enrolling regimen. All participants will have an equal chance of being randomized to any currently enrolling regimen.

If a participant is randomized to Regimen F ABBV-CLS-7262, the participant will complete a screening visit to assess additional Regimen F eligibility criteria.

Once Regimen F eligibility criteria are confirmed, participants will complete a baseline assessment and be randomized in an overall 3:1 ratio to either active ABBV-CLS-7262 or matching placebo. The first 240 participants will be assigned in a 2:1:1 allocation ratio to Dose 1 ABBV-CLS-7262, Dose 2 ABBV-CLS-7262, or placebo. The final approximately 60 participants will be assigned in a 3:1 allocation ratio to Dose 1 ABBV-CLS-7262 or placebo.

Regimen F will enroll by invitation, as participants may not choose to enroll in Regimen F. Participants must first enroll into the Master Protocol and be eligible to participate in the Master Protocol before being able to be randomly assigned to Regimen F.

For a list of enrolling sites, please see the HEALEY ALS Platform Trial Master Protocol under NCT04297683.

ELIGIBILITY:
Inclusion Criteria:

* No additional inclusion criteria beyond the inclusion criteria specified in the Master Protocol (NCT NCT04297683).

Exclusion Criteria:

* The following exclusion criteria are in addition to the exclusion criteria specified in the Master Protocol (NCT NCT04297683).

  1. Based on the metabolism of the compound, the concomitant use of certain inhibitors and inducers of cytochrome P450 enzymes.
  2. Any clinically significant ECG abnormalities.
  3. Clinically significant clinical laboratory abnormalities.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2024-10-03 (Actual); Study Completion 2024-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merit Cudkowicz, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Healey Center for ALS at Mass General, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ABBV-CLS-7262 Dose 1 | ABBV-CLS-7262 Dose 2 | Matching Placebo
Started | 155 | 79 | 76
Completed | 137 | 66 | 71
Not Completed | 18 | 13 | 5

BASELINE CHARACTERISTICS:
Population: Baseline Analysis Population includes only placebo participants from the Regimen F Efficacy Regimen Only (ERO) sample; shared placebo participants from other regimens are not included in the Baseline Analysis Population.
Groups:
- Total: Total of all reporting groups
Arm/Group | ABBV-CLS-7262 Dose 1 | ABBV-CLS-7262 Dose 2 | Matching Placebo | Total
Number analyzed (Participants) | 155 | 79 | 76 | 310
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.3 (11.2) | 58.2 (11.02) | 58.0 (11.13) | 57.7 (11.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 30 | 34 | 124
  Male | 95 | 49 | 42 | 186
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 4 | 1 | 5 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 3 | 6
  White | 145 | 75 | 65 | 285
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 8 | 6 | 26
  Not Hispanic or Latino | 143 | 71 | 70 | 284
  Unknown or Not Reported | 0 | 0 | 0 | 0
ALS Diagnosis from R El Escorial Criteria [Count of Participants; unit: Participants] — The El Escorial Criteria are a set of guidelines used to diagnose ALS based on clinical signs of upper motor neuron and lower motor neuron dysfunction
  Participants
    Clinically Possible ALS | 17 | 7 | 7 | 31
    Clinically Probable ALS - Laboratory Supported | 34 | 10 | 14 | 58
    Clinically Probable ALS | 58 | 28 | 33 | 119
    Clinically Definite ALS | 46 | 34 | 22 | 102
ALS Onset Location [Count of Participants; unit: Participants]
  Axial | 0 | 2 | 0 | 2
  Bulbar | 27 | 8 | 11 | 46
  Generalized | 0 | 1 | 0 | 1
  Limb | 125 | 67 | 65 | 257
  Multiple | 1 | 1 | 0 | 2
  Respiratory | 2 | 0 | 0 | 2
Time Since Symptom Onset at Baseline [Mean (Standard Deviation); unit: Months] | 22.2 (8.07) | 19.6 (7.94) | 19.7 (7.38) | 20.93 (7.95)
Delay in ALS Symptom Onset and Diagnosis [Mean (Standard Deviation); unit: Months] | 10.4 (5.56) | 9.3 (5.44) | 8.9 (4.74) | 9.71 (5.36)
Baseline Edaravone Use [Count of Participants; unit: Participants]
  Yes | 96 | 49 | 46 | 191
  No | 59 | 30 | 30 | 119
Baseline Riluzole Use [Count of Participants; unit: Participants]
  Yes | 133 | 68 | 65 | 266
  No | 22 | 11 | 11 | 44
Baseline Relyvrio Use [Count of Participants; unit: Participants]
  Yes | 90 | 47 | 46 | 183
  No | 65 | 32 | 30 | 127
ALSFRS-R Total Score [Mean (Standard Deviation); unit: Points] — The ALS Functional Rating Score-Revised (ALSFRS-R) measures 12 aspects of physical function. Each of the 12 questions assessing distinct functional ability is scored from 4 (normal) to 0 (no ability), with a maximum total score of 48 and a minimum total score of 0. Participants with higher scores have more physical function.
  Points | 36 (6.54) | 35 (7.67) | 36.8 (6.68) | 35.90 (6.89)
Pre-Baseline Decline in ALSFRS-R [Mean (Standard Deviation); unit: Points per Month] — The pre-baseline decline score is 48-Baseline ALSFRS-R divided by the number of months between onset of weakness due to ALS and the date of Baseline. A higher number indicates faster decline.
  Points per Month | 0.6 (0.44) | 0.8 (0.66) | 0.6 (0.41) | 0.65 (0.51)
SVC [Mean (Standard Deviation); unit: Percent predicted] — Slow vital capacity is an assessment of breathing function. The total amount of air that can be exhaled is measured. A higher slow vital capacity indicates better breathing function.
  Percent predicted | 81.5 (18.31) | 82.0 (17.20) | 85.0 (16.98) | 82.51 (17.72)
King Stage [Count of Participants; unit: Participants] — The King's ALS Clinical Staging System is a 4-level ordinal scale with the first three levels indicating the number (1, 2, or 3) of distinct central nervous system regions (bulbar, upper limb, and lower limb) with neuromuscular dysfunction. Level 4a indicates nutritional failure and level 4b indicates respiratory failure. Higher scores indicate a worse disease state.
  Participants
    1 Region with Neuromuscular Dysfunction | 33 | 18 | 20 | 71
    2 Region with Neuromuscular Dysfunction | 37 | 17 | 20 | 74
    3 Region with Neuromuscular Dysfunction; | 40 | 19 | 22 | 81
    4a/b Nutritional/Respiratory Failure | 45 | 25 | 14 | 84
Weight [Mean (Standard Deviation); unit: Kg] | 82.4 (22.34) | 78.8 (16.68) | 81.1 (19.74) | 81.19 (20.39)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27.4 (6.53) | 26.4 (4.77) | 27.3 (5.33) | 27.12 (5.83)
Serum NfL Concentration [Median (Inter-Quartile Range); unit: ng/L] — Population: Number analyzed in row differs from overall number due to missing data.
  ng/L
    number analyzed (Participants) | 150 | 76 | 69 | 295
    (all) | 52.9 [34.2 to 70.8] | 55.2 [36.2 to 86.4] | 64.4 [36.5 to 91.7] | 54.8 [35.4 to 80.4]
Serum Creatinine Concentration [Mean (Standard Deviation); unit: mg/dL] | 0.7 (0.18) | 0.7 (0.18) | 0.7 (0.20) | 0.7 (0.19)

OUTCOME MEASURES:

1. Primary Outcome: Disease Progression as Assessed by the ALSFRS-R-Slope
Description: Change in disease severity as measured by the ALS Functional Rating Scale-Revised (ALSFRS-R) total score using a Bayesian repeated measures model that accounts for loss to follow-up due to mortality. Each of 12 questions assessing distinct functional ability is scored from 4(normal) to 0 (no ability), with a maximum total score of 48 and a minimum total score of 0. Participants with higher scores have more physical function. Note that only participants who survived to their Week 24 visit contribute to the estimate.
Time Frame: Baseline to 24 Weeks
Population: Outcome measure data was analyzed using the Efficacy Concurrent-controls Set (ECC), which included concurrent shared placebos from other regimens if randomized within 180 days of the first and last randomization for the applicable regimen, excluding any shared placebos also include in the focal regimen, as pre-specified in the Regimen Statistical Analysis Plan. Regimen F (NCT#05740813) and Regimen G (NCT#05842941) contributed placebo participants into the shared placebo cohort used for analysis.
Measure: Mean (Standard Deviation); unit: Points per month
Arm/Group | ABBV-CLS-7262 Dose 1 | ABBV-CLS-7262 Dose 2 | Matching Placebo
Number analyzed (Participants) | 155 | 78 | 126
Points per month | -1.00 (0.068) | -0.91 (0.078) | -0.95 (0.085)
Statistical Analysis 1: Comparison: ABBV-CLS-7262 Dose 1 vs Matching Placebo; Test type: Superiority; Bayesian shared-parameter mode — Posterior probability that the disease rate ratio (DRR) is less than 1 (i.e. ABBV-CLS-7262 slowed progression) was 0.3117 for Dose 1. NOTE: p-value is not provided for Bayesian model; A Bayesian shared-parameter model of change in disease severity as measured by ALSFRS-R total score and mortality; Disease Rate Ratio = 1.06, 95% CI 2-sided [0.850 to 1.324], Standard Deviation 0.120 — DDR <1 imply slowing of disease progression by ABBV-CLS-7262 relative to placebo. Note: reported "Confidence Interval" is actually a Bayesian credible interval; The DRR parameter for active treatment represents the relative change to the rate of decline of ALSFRS-R and the rate of mortality of treated participant relative to a placebo participant. The estimated DRR can also be interpreted as the average rate of decline in function and mortality. The model incorporates participant-level random effects in the baseline value of the ALSFRS-R (intercept) and in the rate of progression (slope); covariate effects to account for covariate-explainable differences in rates of progression based on participant-specific baseline covariates; regimen-specific differences in baseline values, rates of progression and measurement error. Covariates include time since onset of symptoms, pre-baseline slope of ALSFRS-R, riluzole, edaravone, and Relyvrio use at the time of baseline as indicated in concomitant medication logs, and log-transformed baseline serum NfL
Statistical Analysis 2: Comparison: ABBV-CLS-7262 Dose 2 vs Matching Placebo; Test type: Superiority; Bayesian shared-parameter model — Posterior probability that the disease rate ratio (DRR) is less than 1 (i.e. ABBV-CLS-7262 slowed progression) was 0.6426. NOTE: p-value is not provided for Bayesian model; A Bayesian shared-parameter model of change in disease severity as measured by ALSFRS-R total score and mortality; Disease Rate Ratio = 0.96, 95% CI 2-sided [0.753 to 1.220], Standard Deviation 0.119 — [estimate comment as in outcome 1, analysis 1]; [other analysis details as in outcome 1, analysis 1]

2. Secondary Outcome: Function by ALSFRS-R Total Score
Description: Change from baseline to Week 24 in function as assessed by ALSFRS-R total score.
Time Frame: Baseline to 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Points
Arm/Group | ABBV-CLS-7262 Dose 1 | ABBV-CLS-7262 Dose 2 | Matching Placebo
Number analyzed (Participants) | 155 | 78 | 126
Points | -6.110 (0.3710) | -5.468 (0.5252) | -5.563 (0.4106)
Statistical Analysis 1: Comparison: ABBV-CLS-7262 Dose 1 vs Matching Placebo; Test type: Superiority; p = 0.3325, Mixed Models Analysis; Covariates: baseline (BL) use edaravone, riluzole, Relyvrio, BL log-trans. NfL, SVC, time since onset, pre-BL ALSFRS-R slope, interactions with visit; Mean Difference (Net) = -0.547, 95% CI 2-sided [-1.657 to 0.562], Standard Error of Mean 0.5639 — ABBV-CLS-7262 Dose 1 24-week change from baseline relative to placebo 24-week change from baseline; Model adjusted for covariates including baseline (BL) use of edaravone, riluzole and Relyvrio, BL log-transformed NfL, and SVC, time since onset, pre-BL ALSFRS-R slope and interaction with visit
Statistical Analysis 2: Comparison: ABBV-CLS-7262 Dose 2 vs Matching Placebo; Test type: Superiority; p = 0.8878, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 0.095, 95% CI 2-sided [-1.230 to 1.420], Standard Error of Mean 0.6732 — ABBV-CLS-7262 Dose 2 24-week change from baseline relative to placebo 24-week change from baseline; [other analysis details as in outcome 2, analysis 1]

3. Secondary Outcome: Respiratory Function
Description: Change in respiratory function over time as measured by Slow Vital Capacity (SVC).
Time Frame: Baseline to 24 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: 24-week diff. of percents of normal VC
Arm/Group | ABBV-CLS-7262 Dose 1 | ABBV-CLS-7262 Dose 2 | Matching Placebo
Number analyzed (Participants) | 155 | 78 | 126
24-week diff. of percents of normal VC | -10.882 (1.3311) | -7.202 (1.9469) | -9.462 (1.5259)
Statistical Analysis 1: Comparison: ABBV-CLS-7262 Dose 1 vs Matching Placebo; Test type: Superiority; p = 0.5008, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -1.420, 95% CI 2-sided [-5.563 to 2.723], Standard Error of Mean 2.1066 — ABBV-CLS-7262 Dose 1 24-week change from baseline relative to placebo 24-week change from baseline; [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: ABBV-CLS-7262 Dose 2 vs Matching Placebo; Test type: Superiority; p = 0.3721, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 2.261, 95% CI 2-sided [-2.714 to 7.236], Standard Error of Mean 2.5292 — ABBV-CLS-7262 Dose 2 24-week change from baseline relative to placebo 24-week change from baseline; [other analysis details as in outcome 2, analysis 1]

4. Primary Outcome: Mortality Event Rate
Description: Mortality is defined as death or death equivalent. A participant is determined to meet the criteria of death equivalent if permanent assisted ventilation (PAV) is used for more than 22 hours per day for more than seven days in a row. The rate of mortality was estimated from a Bayesian shared-parametric model that assumed exponentially distributed survival times.
Time Frame: Baseline to 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Events per month
Arm/Group | ABBV-CLS-7262 Dose 1 | ABBV-CLS-7262 Dose 2 | Matching Placebo
Number analyzed (Participants) | 155 | 78 | 126
Events per month | 0.009 (0.0022) | 0.008 (0.0021) | 0.009 (0.0022)

5. Secondary Outcome: Upper Limb Muscle Strength
Description: Change in upper limb muscle strength over time as measured isometrically using hand-held dynamometry and grip strength, calculated as the average percent change from baseline of the following muscles/maneuvers: shoulder flexion, elbow flexion, elbow extension, wrist extension, abductor pollicis brevis contraction, abductor digiti minimi contraction, first dorsal interosseous contraction, and grip strength. Note that only those with measurable strength at baseline were included.
Time Frame: Baseline to 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | ABBV-CLS-7262 Dose 1 | ABBV-CLS-7262 Dose 2 | Matching Placebo
Number analyzed (Participants) | 155 | 78 | 126
Percent change | -36.281 (2.6896) | -25.760 (3.8365) | -38.078 (3.0500)
Statistical Analysis 1: Comparison: ABBV-CLS-7262 Dose 1 vs Matching Placebo; Test type: Superiority; p = 0.6707, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 1.796, 95% CI 2-sided [-6.506 to 10.099], Standard Error of Mean 4.2220 — ABBV-CLS-7262 Dose 1 24-week change from baseline relative to placebo 24-week change from baseline; [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: ABBV-CLS-7262 Dose 2 vs Matching Placebo; Test type: Superiority; p = 0.0144, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 12.318, 95% CI 2-sided [2.463 to 22.172], Standard Error of Mean 5.0110 — ABBV-CLS-7262 Dose 2 24-week change from baseline relative to placebo 24-week change from baseline; [other analysis details as in outcome 2, analysis 1]

6. Secondary Outcome: Disease Progression Biomarker
Description: Change in log-transformed serum neurofilament light protein (NfL) concentration from baseline to Week 24.
Time Frame: Baseline to 24 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ln(ng/L)
Arm/Group | ABBV-CLS-7262 Dose 1 | ABBV-CLS-7262 Dose 2 | Matching Placebo
Number analyzed (Participants) | 155 | 78 | 126
ln(ng/L) | 0.086 (0.0247) [1.038 to 1.144] | 0.067 (0.0355) [0.997 to 1.146] | -0.002 (0.0282) [0.944 to 1.055]
Statistical Analysis 1: Comparison: ABBV-CLS-7262 Dose 1 vs Matching Placebo; Test type: Superiority; p = 0.0253, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 1.092, 95% CI 2-sided [1.011 to 1.179] — Least squares mean difference between ABBV-CLS-7262 Dose 1 24-week change from baseline and placebo 24-week change from baseline; Model adjusted for covariates including baseline (BL) use of edaravone, riluzole and Relyvrio, BL log-transformed NfL, SVC, time since onset, pre-BL ALSFRS-R slope and interaction with visit
Statistical Analysis 2: Comparison: ABBV-CLS-7262 Dose 2 vs Matching Placebo; Test type: Superiority; p = 0.1364, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 1.073, 95% CI 2-sided [0.978 to 1.175] — Least squares mean difference between ABBV-CLS-7262 Dose 2 24-week change from baseline and placebo 24-week change from baseline; [other analysis details as in outcome 6, analysis 1]

7. Secondary Outcome: Activities of Daily Living
Description: Change from baseline to Week 24 in the activities of daily living (ADL)/independence domain score as assessed by the Amyotrophic Lateral Sclerosis Assessment Questionnaire-40 (ALSAQ-40). The ALSAQ-40, a patient-self reported outcome, consists of 40 questions that are used to measure the subjective well-being of participants, and each question is scored from 0 (never) to 5 (always or cannot do at all). The ADL/independence domain score is based on 10 out of the 40 questions, with a maximum ADL/independence domain score of 50 and minimum score of 0. Higher domain scores indicate a worse subjective well-being or less independence completing ADLs.
Time Frame: Baseline to 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Points
Arm/Group | ABBV-CLS-7262 Dose 1 | ABBV-CLS-7262 Dose 2 | Matching Placebo
Number analyzed (Participants) | 155 | 78 | 126
Points | 13.643 (1.2961) | 12.049 (1.8617) | 13.701 (1.5115)
Statistical Analysis 1: Comparison: ABBV-CLS-7262 Dose 1 vs Matching Placebo; Test type: Superiority; p = 0.9782, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -0.058, 95% CI 2-sided [-4.254 to 4.137], Standard Error of Mean 2.1327 — ABBV-CLS-7262 Dose 1 24-week change from baseline relative to placebo 24-week change from baseline; [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: ABBV-CLS-7262 Dose 2 vs Matching Placebo; Test type: Superiority; p = 0.5108, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -1.652, 95% CI 2-sided [-6.590 to 3.286], Standard Error of Mean 2.5101 — ABBV-CLS-7262 Dose 2 24-week change from baseline relative to placebo 24-week change from baseline; [other analysis details as in outcome 2, analysis 1]

8. Secondary Outcome: Number of Participants That Experienced Death or Death Equivalent
Description: The number of participants who died or met the criterion for a death equivalent from the date of their baseline visit to the end of the Week 24visit window (generally 175 days after baseline). The death equivalent criterion is use of permanent assisted ventilation (PAV) for more than 22 hours per day for more than 7 days in a row.
Time Frame: Baseline to 24 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ABBV-CLS-7262 Dose 1 | ABBV-CLS-7262 Dose 2 | Matching Placebo
Number analyzed (Participants) | 155 | 79 | 126
Participants | 8 | 4 | 5
Statistical Analysis 1: Comparison: ABBV-CLS-7262 Dose 1 vs Matching Placebo; Test type: Superiority; p = 0.6481, Log Rank; Dose 1. See Other Statistical Analysis for model adjustment details; Cox proportional hazards model adjusted for age at baseline, time since ALS symptom onset, delta FRS, baseline log-transformed serum NfL level, use of riluzole at baseline, use of riluzole at baseline, and use of Relyvrio at baseline
Statistical Analysis 2: Comparison: ABBV-CLS-7262 Dose 2 vs Matching Placebo; Test type: Superiority; p = 0.6344, Log Rank; Dose 2. See Other Statistical Analysis for model adjustment details; [other analysis details as in outcome 8, analysis 1]

ADVERSE EVENTS:
Time Frame: Up to 35 weeks after participant signed Master Protocol consent
Arm/Group | ABBV-CLS-7262 Dose 1 | ABBV-CLS-7262 Dose 2 | Matching Placebo
All-Cause Mortality (participants affected / at risk) | 6/155 | 3/79 | 1/76
Serious Adverse Events (participants affected / at risk) | 21/155 | 7/79 | 6/76
Other Adverse Events (participants affected / at risk) | 125/155 | 59/79 | 62/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABBV-CLS-7262 Dose 1 (N=155) | ABBV-CLS-7262 Dose 2 (N=79) | Matching Placebo (N=76)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Complication associated with device (General disorders) | 1 (1) | 1 (1) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Acinetobacter bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 2 (3) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Traumatic intracranial haematoma (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasticity (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Muscular weakness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Device malfunction (Product Issues) | 2 (2) | 0 (0) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0)
Cardio-respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABBV-CLS-7262 Dose 1 (N=155) | ABBV-CLS-7262 Dose 2 (N=79) | Matching Placebo (N=76)
Abdominal pain (Gastrointestinal disorders) | 9 (9) | 5 (5) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 4 (5) | 0 (0)
Constipation (Gastrointestinal disorders) | 23 (24) | 10 (12) | 12 (12)
Diarrhoea (Gastrointestinal disorders) | 17 (18) | 9 (10) | 8 (11)
Dysphagia (Gastrointestinal disorders) | 5 (6) | 5 (6) | 6 (6)
Nausea (Gastrointestinal disorders) | 10 (11) | 3 (3) | 4 (6)
Salivary hypersecretion (Gastrointestinal disorders) | 11 (11) | 7 (7) | 4 (4)
Fatigue (General disorders) | 9 (10) | 6 (6) | 7 (8)
COVID-19 (Infections and infestations) | 13 (13) | 6 (6) | 4 (4)
Nasopharyngitis (Infections and infestations) | 8 (9) | 6 (6) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 3 (3) | 6 (6)
Urinary tract infection (Infections and infestations) | 6 (7) | 6 (7) | 4 (7)
Contusion (Injury, poisoning and procedural complications) | 4 (4) | 7 (12) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 47 (83) | 28 (72) | 31 (69)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 12 (13) | 8 (9) | 8 (9)
Post-traumatic pain (Injury, poisoning and procedural complications) | 2 (2) | 2 (4) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 4 (6) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 6 (7) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (5) | 2 (2)
Cognitive disorder (Nervous system disorders) | 6 (6) | 1 (1) | 4 (4)
Dizziness (Nervous system disorders) | 11 (14) | 1 (1) | 10 (13)
Dysarthria (Nervous system disorders) | 6 (6) | 4 (4) | 5 (5)
Headache (Nervous system disorders) | 21 (23) | 9 (9) | 12 (15)
Muscle contractions involuntary (Nervous system disorders) | 2 (2) | 3 (3) | 4 (6)
Muscular weakness (Nervous system disorders) | 19 (32) | 13 (21) | 14 (28)
Neuromyopathy (Nervous system disorders) | 11 (16) | 13 (20) | 8 (9)
Anxiety (Psychiatric disorders) | 3 (3) | 6 (7) | 4 (4)
Depression (Psychiatric disorders) | 2 (2) | 4 (5) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 4 (4) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 7 (7) | 8 (9)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 9 (9) | 2 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-07-23): https://cdn.clinicaltrials.gov/large-docs/13/NCT05740813/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-13): https://cdn.clinicaltrials.gov/large-docs/13/NCT05740813/SAP_001.pdf